CLINICAL TRIAL: NCT05523778
Title: A Multi-center Study to Evaluate the Efficacy and Safety of Pancreatic Duct Stents Placement Before the Enucleation of Insulinoma Located in the Head and Neck of the Pancreas Near the Main Pancreatic Duct
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University First Hospital (Other); Xuanwu Hospital, Beijing (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PANCSTENTEN
Record Dates: First submitted 2022-08-16; First posted 2022-08-31 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-07

CONDITIONS: Insulinoma
Keywords: Pancreatic enucleation; Pancreatic duct stent; Regular pancreatectomy; Health economics evaluation
MeSH Terms: conditions — Insulinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are kept blinded to participant group allocation. Objective clinical data are provided to independent assessors with blindness of allocation. With clear definition for each endpoints, assessors are able to make grading for complications in primary and secondary endpoints
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stented EN (Experimental): Patients are placed the pancreatic duct stent by endoscopist 1day or several hours before the enucleation surgery.
  Interventions: Procedure: placement of pancreatic duct stents before enucleation surgery
- Direct EN (Active Comparator): Patients will receive enucleation surgery directly following normal procedure
  Interventions: Procedure: Direct enucleation surgery

INTERVENTIONS:
Procedure: placement of pancreatic duct stents before enucleation surgery — Advance placement of pancreatic stents endoscopically
  Arms: Stented EN
Procedure: Direct enucleation surgery — Patients will receive direct enucleation surgery
  Arms: Direct EN

SUMMARY:
The purpose of this study is to compare the clinical efficacy and economic cost of enucleation after placement of pancreatic duct stents before surgery with that of direct enucleation alone, and to evaluate its safety and feasibility.

DETAILED DESCRIPTION:
The research contents of this study include: patients with insulinoma near the main pancreatic duct in the head and neck of the pancreas were randomly divided into two groups: the preoperative pancreatic duct stent enucleation group (stended EN), the direct en group (DEN), the Sen group asked a digestive endoscopist to place the pancreatic duct stent before surgery, and the next day or the next day after surgery, and the den group received enucleation directly. The safety of the two groups was compared, including the evaluation of surgical effect Postoperative complications and long-term prognosis based on follow-up data analysis; At the same time, the differences between the two groups were evaluated from the perspective of health economics.

ELIGIBILITY:
Inclusion Criteria:

* The clinical qualitative diagnosis of insulinoma was clear;
* The localization diagnosis was clear, and it was determined that the tumor was single, located in the head and neck;
* The distance between the tumor and the main pancreatic duct was determined to be ≤ 2mm by preoperative imaging (enhanced CT, MRI, etc.);
* Truly informed and voluntarily participate in this study.

Exclusion Criteria:

* Maximum diameter of the tumor >2cm proved pathologically
* Severe cardiopulmonary complications before operation
* Combined with other known tumor diseases
* Insulinoma is invasive or has suspicious metastatic lesions
* Previous upper abdominal surgery history
* Refusal or inability to cooperate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of POPF within 3 months after EN. | 3 days to 3 months after enucleation (or the extubation time),up to 6 month after inclusion
  Postoperative clinically relevant pancreatic fistula in this study adopts the definition proposed by the international pancreatic surgery research group (ISGPS)

SECONDARY OUTCOMES:
Rate of postoperative abdominal infection within 3 weeks after EN | 3 days to 3 weeks after enucleation (or the extubation time),,up to 6 month after inclusion
  Abdominal infection can be basically diagnosed if one of the following conditions occurs:
  1. After 3 days of operation, the patient developed chills, high fever, abdominal distension, intestinal paralysis, etc., which lasted for more than 24 hours. The laboratory examination results showed that the leukocyte count increased significantly, with or without hypoproteinemia and anemia, and the imaging images showed the accumulation of fluid in the abdominal cavity;
  2. The aspiration fluid was purulent or bacteria were detected in the fluid;
  3. The infection was localized and formed inclusion. In imaging, fluid accumulation foci with clear edges and with or without gas could be seen.
Rate of postoperative delayed gastric emptying within 3 weeks after EN | 3 days to 3 weeks after enucleation (or the extubation time)
  Gastric emptying disorder can be diagnosed if the solid diet cannot be restored 1 week after operation and the gastric tube cannot be removed.
Rate of postoperative hemorrhagepostpancreatectomy haemorrhage within 3 weeks after EN | 1 days to 3 weeks after enucleation (or the extubation time),,up to 6 month after inclusion
  Postoperative hemorrhage refers to the occurrence of bloody fluid in the abdominal drainage tube or gastrointestinal decompression tube, which can also be manifested as blood in the stool, accompanied by changes in vital signs such as heart rate and blood pressure, as well as a decrease in hemoglobin concentration.
Rate of postoperative dyspepsia within 6 months after EN | 2 weeks to 6 months after enucleation,,up to 6 month after inclusion
  According to Rome IV standard, the diagnosis should meet the following requirements:
  Symptoms appear for at least 2 months, and must include one or more of the following uncomfortable symptoms, and at least 4 times a month:
  a. fullness after meals; b. Early satiety; c. Epigastric pain or burning sensation has nothing to do with defecation; d. After proper evaluation, the symptoms cannot be completely explained by other disease conditions.
Rate of postoperative lung infection within 3 weeks after EN | 1 days to 3 weeks after enucleation (or the extubation time),,up to 6 month after inclusion
  Patients with any of the following conditions:
  a. continuous fever or leukocytosis, accompanied by postoperative chest X-ray or chest CT positive findings (consolidation of lung, pneumonia, atelectasis, with or without pleural effusion), and decreased body temperature after antibiotics; b. Sputum culture is positive, accompanied by continuous fever or leukocyte elevation, and body temperature drops after antibiotics; c. Pleural effusion affects the patient's breathing and requires pleural puncture and drainage.
Rate of postoperative hyperglycemia within 6 months after EN | 2 weeks to 6 months after enucleation,,up to 6 month after inclusion
  the diagnosis should meet at least one of the following requirements:
  a. hemoglobin A1c (HbA1c) value ≥ 6.5%; b. If the fasting blood glucose is ≥ 126mg / dl, the test should be repeated on another day. Fasting is defined as at least 8 hours without calorie intake; c. Oral glucose tolerance test (OGTT), plasma glucose ≥ 200 mg / dl at 2 hours after 75g (100g for pregnant women) glucose load; d. Hyperglycemic symptoms and accidental (random) plasma glucose ≥ 200mg / dl.
Rate of post-stent-placement acute pancreatitis in Stented EN group within in 3 weeks after EN | 1 days to 3 days after stent placement,,up to 6 month after inclusion
  Patients with any two of the following three criteria can be diagnosed : a. abdominal pain consistent with the onset; b. Biochemical evidence of pancreatitis (serum amylase and / or lipase greater than 3 times the upper limit of normal); c. Typical manifestations of abdominal image (pancreatic edema / necrosis or exudation and effusion around the pancreas)
Operation time | Measure during operation,,up to 6 month after inclusion
Intraoperative blood loss | Measure during operation,,up to 6 month after inclusion
Total cost of hospitalization | Measure during the whole hospitalization procedure of each patient,,up to 6 month after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in the surgical treatment of insulinoma. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis."Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Gao R, Yin B, Jin J, Tian X, Zhang Y, Wei J, Cao F, Wang Z, Ma Z, Wang M, Gou S, Cong L, Xu Q, Wu W, Zhao Y. Preoperative pancreatic stent placement before the enucleation of insulinoma located in the head and neck of the pancreas in proximity to the main pancreatic duct: study protocol for a multicentre randomised clinical trial in Chinese tertiary medical centres. BMJ Open. 2024 Apr 2;14(4):e078516. doi: 10.1136/bmjopen-2023-078516. PMID 38569703